CLINICAL TRIAL: NCT00738946
Title: A Trial of the Combined Impact of Intermittent Preventive Treatment and Insecticide Treated Bednets in Reducing Morbidity From Malaria in African Children
Acronym: IPTc/ITNs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Centre national de recherche et de formation sur le paludisme (Other Government); Malaria Research and Training Centre, Mali (Unknown)
Responsible Party: Professor Brian Greenwood, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IPTCVP17; NCT00745979 (obsolete NCT alias)
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-06

CONDITIONS: Malaria
Keywords: Intermittent Preventive treatment; insecticide treated bednets; malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Experimental): Amodiaquine+pyrimethamine versus placebo
  Interventions: Drug: Intermittent preventive treatment with AQ+ SP

INTERVENTIONS:
Drug: Intermittent preventive treatment with AQ+ SP — Amodiaquine (10 mg/kg over 3 days) and Sulfadoxine Pyrimethamine (25 mg of sulfadoxine + 1.25 mg of pyrimethamine per kg in a single dose) or placebo administered over 3 rounds of one month interval
  Other Names: IPTc

SUMMARY:
An investigation will be made of the combined impact of insecticide-treated nets and intermittent preventive treatment with amodiaquine + sulfadoxine-pyrimethamine on malaria morbidity in children in Burkina Faso and Mali.Three rounds of treatment will be given during the malaria season in one year and the follow-up will be extended into the second year by passive surveillance.

DETAILED DESCRIPTION:
The trial will be conducted in 6000 children in Burkina Faso and Mali in 2008 and 2009. Each site will enroll 3,000 children. All children will be allocated a long lasting insecticide-treated net and randomized to receive to treatment (amodiaquine + sulfadoxine-pyrimethamine (AQ+SP)) or placebo (AQ-placebo + SP-placebo. Treatment will be administered over 3 rounds during the high malaria transmission season, with one month interval between rounds. Full course treatment of AQ and SP will be administered on each occasion. Treatment will not be given in the second year. Passive surveillance of malaria will be implemented for the monitoring of malaria morbidity and to assess whether children who received intermittent preventive treatment (IPT) are at increased risk of malaria. Adverse events will be monitored during each round of IPT administration. To assess the effect of IPTc on the prevalence of malaria infection, a random sample of 150 children will be visited every week during the high malaria transmission period. This number will be increased to 300 during the low transmission season, but the survey will be reduced to monthly visits. Baseline prevalence of genetic markers of resistance to SP and AQ will be estimated. A second cross-sectional survey will be conducted at the end of the malaria transmission season to assess the effect of IPT on the prevalence of genetic markers of resistance to SP and AQ, on the prevalence of anaemia and on nutritional indicators.

ELIGIBILITY:
Inclusion Criteria:

* Permanent residence in the study area with no intention of leaving during the surveillance period.
* Obtention of informed consent.

Exclusion Criteria:

* Temporary residence in the study area.
* Absence of informed consent.
* Presence of a severe, chronic illness such as severe malnutrition (Kwashiorkor or marasmus) or AIDS, likely to interfere with evaluation of the trial results.
* A history of a previous, significant adverse reaction to either of the study drugs.

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6000 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Incidence of clinical malaria | 2008-2009

SECONDARY OUTCOMES:
Incidence of severe malaria, Incidence of anemia, Prevalence of anemia, Prevalence of parasitemia, Proportion of children with parasites carrying resistance markers to AQ and SP, Incidence of hospital admissions due to malaria. | 2008-2009

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Greenwood, MD, FRCP, Study Director — London School of Hygiene and Tropical Medicine
Locations (2):
- Centre National de Recherche et de Formation sur le Paludisme, Ouagadougou, Kadiogo, Burkina Faso
- Malaria Research and Training Centre, Bamako, Mali

REFERENCES:
- [Derived] Konate AT, Yaro JB, Ouedraogo AZ, Diarra A, Gansane A, Soulama I, Kangoye DT, Kabore Y, Ouedraogo E, Ouedraogo A, Tiono AB, Ouedraogo IN, Chandramohan D, Cousens S, Milligan PJ, Sirima SB, Greenwood BM, Diallo DA. Morbidity from malaria in children in the year after they had received intermittent preventive treatment of malaria: a randomised trial. PLoS One. 2011;6(8):e23391. doi: 10.1371/journal.pone.0023391. Epub 2011 Aug 12. PMID 21858097
- [Derived] Dicko A, Barry A, Dicko M, Diallo AI, Tembine I, Dicko Y, Dara N, Sidibe Y, Santara G, Conare T, Chandramohan D, Cousens S, Milligan PJ, Diallo DA, Doumbo OK, Greenwood B. Malaria morbidity in children in the year after they had received intermittent preventive treatment of malaria in Mali: a randomized control trial. PLoS One. 2011;6(8):e23390. doi: 10.1371/journal.pone.0023390. Epub 2011 Aug 12. PMID 21858096
- [Derived] Konate AT, Yaro JB, Ouedraogo AZ, Diarra A, Gansane A, Soulama I, Kangoye DT, Kabore Y, Ouedraogo E, Ouedraogo A, Tiono AB, Ouedraogo IN, Chandramohan D, Cousens S, Milligan PJ, Sirima SB, Greenwood B, Diallo DA. Intermittent preventive treatment of malaria provides substantial protection against malaria in children already protected by an insecticide-treated bednet in Burkina Faso: a randomised, double-blind, placebo-controlled trial. PLoS Med. 2011 Feb 1;8(2):e1000408. doi: 10.1371/journal.pmed.1000408. PMID 21304925
- [Derived] Dicko A, Diallo AI, Tembine I, Dicko Y, Dara N, Sidibe Y, Santara G, Diawara H, Conare T, Djimde A, Chandramohan D, Cousens S, Milligan PJ, Diallo DA, Doumbo OK, Greenwood B. Intermittent preventive treatment of malaria provides substantial protection against malaria in children already protected by an insecticide-treated bednet in Mali: a randomised, double-blind, placebo-controlled trial. PLoS Med. 2011 Feb 1;8(2):e1000407. doi: 10.1371/journal.pmed.1000407. PMID 21304923